CLINICAL TRIAL: NCT06569875
Title: Feasibility Study: Self-guided Internet-based Cognitive Behavioral Therapy as a Stepped-care Treatment for Mothers With Postpartum Depression.
Brief Title: Feasibility Study: Self-guided iCBT for Mothers With Postpartum Depression.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other); University of Copenhagen (Other); University of Aarhus (Other)
Responsible Party: Principal Investigator, Trine Munk-Olsen, Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12.250
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Postpartum Depression; Internet-based Intervention
Keywords: Cognitive behavioral therapy; Postpartum depression; Web-based intervention
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based cognitive behavioural therapy program (Experimental): Participants will have access to an internet-based cognitive behavioral therapy program called iCARE for eight weeks.
  Interventions: Device: iCARE
- Treatment as usual (No Intervention): Participants in the control group will receive treatment as usual in their municipality.

INTERVENTIONS:
Device: iCARE — iCARE is an internet-based cognitive behavioral therapy program designed for women experiencing symptoms of postpartum depression, including anxiety, irritability, and sadness. The program offers digital therapy through an online platform tailored to mothers with mild to moderate postpartum depression. The program consists of 7 modules, each with its own theme, incorporating cognitive behavioral therapy, a well-established therapeutic approach for depression. The content includes text, images, audio files, and short films, supplemented with small tasks to provide knowledge and tools to understand and manage one's situation. The treatment course is self-directed, allowing participants to engage with the content at their own pace and at times that are most convenient for them
  Arms: Internet-based cognitive behavioural therapy program

SUMMARY:
The purpose of this study is to conduct a feasibility study to test the study procedure and a newly developed self-guided internet-based cognitive behavioral therapy program for mothers with postpartum depression.

DETAILED DESCRIPTION:
The aim of the feasibility study is twofold: 1) to test the feasibility of the study, and 2) to test the acceptability of the internet-based cognitive behavioral therapy program and to minimize dropout.

The study will be conducted as a mixed-method process evaluation. Twenty mothers will be included in the study. After being informed about the study and its potential, all patients who give written informed consent will be randomized in a 1:1 ratio into either the control group, receiving treatment as usual, or the intervention group, receiving treatment as usual plus the iCBT program iCARE. The intervention period will last for two months.

After the intervention period, investigators will use a survey distributed from REDCap to measure its feasibility, participants' satisfaction with it, and acceptability.

After the two-month intervention period, semi-structured interviews will be conducted with participants from both the intervention and control groups to gather qualitative insights. This feasibility study will also provide a preliminary evaluation of the intervention's impact. The findings from this pilot study will inform the design of the subsequent randomized controlled trial (RCT) and guide any necessary modifications to the treatment program and associated procedures.

ELIGIBILITY:
Inclusion Criteria:

* Edinburgh Postnatal Depression Scale (EPDS) score 11-18
* ≥age 18
* Access to the internet

Exclusion Criteria:

* Thoughts of self-harm≥2 on EPDS item 10
* Do not understand Danish language,
* Substance abuse or dependence
* Alcohol abuse, defined as a weekly consumption of alcohol exceeding ten units,
* Physical condition requiring frequent hospitalization like dialysis, chemotherapy, or blood transfusion,
* A diagnosis of schizophrenia or other psychotic disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
The feasibility of the trial procedure will be assessed as a composite outcome consisting of: | Baseline, two-month follow-up, and the six-month follow-up
  * Data collection feasibility: measured as assessment completion
  * Recruitment: measured as the total number of eligible participants, the number who completed the screening questionnaire, and the number of participants completing enrollment per month
  * Experiences with the trial procedures: Post-intervention, all enrolled participants will participate in a semi-structured interview to evaluate their experiences with the trial procedures. A member of the research team will conduct the interviews.

SECONDARY OUTCOMES:
The acceptability of the intervention will be assessed as a composite outcome consisting of: | Two-month follow-up
  The acceptability of the intervention will be assessed as a composite outcome consisting of:
  * The Client Satisfaction Questionnaire (CSQ-8) will measure participants' satisfaction with the intervention. The questionnaire consists of eight items measured on a four-point scale, with total scores ranging from 8 to 32, with a higher number indicating greater satisfaction.
  * The System Usability Scale (SUS) will measure participants' perceptions of the software's usability. The questionnaire consists of ten items measured on a five-point scale, with total scores ranging from 0 to 100, with a higher number indicating a better outcome.
  * Experiences using the intervention: Post-intervention, participants in the intervention group will assess their experiences using the intervention and any issues related to it. A research team member will conduct semi-structured interviews with the participants.

OTHER OUTCOMES:
Severity of depressive symptoms | Baseline, two-month follow-up, and the six-month follow-up
  Edinburg Postnatal Depression Scale (EPDS). It is a ten-item questionnaire, with scores ranging from 0 to 30. Higher scores indicate a worse outcome.
Adverse effects of the intervention | Two-month follow-up
  Negative Effects Questionnaire (NEQ). The questionnaire includes general information about the possibility of experiencing negative effects and is comprised of three separate parts: 1) "Did you experience this?" (yes/no) 2) "If yes-here is how negatively it affected me" (not at all, slightly, moderately, very, and extremely), and 3) "Probably caused by" (the treatment I received/other circumstances). The questionnaire contains 32 items, and how negatively the negative effect was is measured on a four-point Likert scale, ranging from 0-4 ("0" being minimum and "4" being maximum). Higher scores indicate a worse outcome.
The frequency of occurrence of automatic negative thoughts | Two-month follow-up
  The Automatic Thoughts Questionnaire (ATQ). The questionnaire consists of 30 items with a 5-point Likert scale. Scores range from 30 to 150, with higher scores indicating a worse outcome.
Individuals' typical levels of difficulties in emotion regulation | Two-month follow-up
  The Difficulties in Emotion Regulation Scale - 16-item version (DERS-16). The questionnaire consists of 16 items that assess emotion regulation difficulties. The total score ranges from 16 to 80, with higher scores indicating more difficulties with emotion regulation.
Level of stress associated with raising children | Two-month follow-up
  Danish Parental Stress Scale (DPSS). This is an 18-item measure of parental stress rated on a five-point scale (Strongly disagree, Disagree, Undecided, Agree, Strongly agree). The total score range is from 18 to 90, and a low score indicates less stress.
The social-emotional development of children | Two-month follow-up
  The Ages and Stages Questionnaire Social-Emotional Six Month (ASQ-SE-2): The questionnaire comprises 23 scored items with higher scores indicating a worse outcome.
Disability/functioning | Baseline, two-month follow-up, and the six-month follow-up
  World Health Organization disability assessment schedule 2.0 12 items: The questionnaire consists of 12 items, measured by a 5-point scale, with scores ranging from 12 to 60. Higher scores indicate a worse outcome.
levels of anxiety | Baseline, two-month follow-up, and the six-month follow-up
  Generalized Anxiety Disorder Assessment (GAD-7): This questionnaire screens levels of anxiety and consists of 7 items scored on a 0-3 scale from 0 to 21. Higher scores indicate a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Trine Munk-Olsen, prof., Principal Investigator — University of Southern Denmark

IPD SHARING:
Plan to Share IPD: No